CLINICAL TRIAL: NCT03940118
Title: A Randomized Study on the Safety and Tolerability of Mechanical Insufflation-exsufflation and Hypertonic Saline With Hyaluronic Acid for Suctioning of Respiratory Tract Secretions in Patients With Artificial Airway
Brief Title: Safety of Mechanical Insufflation-exsufflation and Hypertonic Saline
Acronym: SMASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Chiesi España (Unknown); Philips Respironics (Industry)
Responsible Party: Principal Investigator, Miguel Sanchez Garcia, Director Critical Care. MD. PhD., Hospital San Carlos, Madrid
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 18/253-R_X
Record Dates: First submitted 2018-12-30; First posted 2019-05-07 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Endotracheal Tube; Tracheostomy
Keywords: respiratory secretion suctioning; mechanical insufflation exsufflation; hypertonic saline; hyaluronic acid; critically ill; artificial airway
MeSH Terms: conditions — Critical Illness | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Intervention Model Description: Randomized, four groups of different respiratory tract secretion suctioning methods: 1) catheter (conventional), 2) catheter after hypertonic saline, 3) mechanical insufflation-exsufflation, and 4) mechanical insufflation-exsufflation with hypertonic saline
Who Masked: Investigator
Masking Description: Closed envelop to be opened after inclusion/exclusion criteria are met and informed consent obtained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Catheter secretion suctioning (Active Comparator): Secretions are aspirated with a catheter at -120 to -150 mBar
  Interventions: Device: Catheter secretion suctioning
- Secretion suctioning + hypertonic saline (Experimental): Hypertonic saline is nebulized prior to aspiration of secretions.
  Interventions: Combination Product: Secretion suctioning + hypertonic saline
- Ins-exsufflation (Experimental): Mechanical insufflation-exsufflation with device programmed at 50/-50 mmHg
  Interventions: Device: Ins-exsufflation
- Ins-exsufflation + Hypertonic Saline (Experimental): Mechanical insufflation-exsufflation and hypertonic saline
  Interventions: Combination Product: Ins-exsufflation + Hypertonic saline

INTERVENTIONS:
Device: Catheter secretion suctioning — Catheter secretion suctioning with prior nebulization of hypertonic saline
  Arms: Catheter secretion suctioning
Combination Product: Secretion suctioning + hypertonic saline — Catheter secretion suctioning with prior nebulization of hypertonic saline
  Arms: Secretion suctioning + hypertonic saline
Device: Ins-exsufflation — Application of a mechanical insufflation-exsufflation device for respiratory tract secretion suctioning
  Arms: Ins-exsufflation
Combination Product: Ins-exsufflation + Hypertonic saline — Application of a mechanical insufflation-exsufflation device for respiratory tract secretion suctioning
  Arms: Ins-exsufflation + Hypertonic Saline

SUMMARY:
Conventional catheter suctioning of respiratory tract secretions is a mandatory procedure in intubated patients. Poor tolerance, pain and other, sometimes severe, lung and cardiovascular complications may occur during suctioning.

Mechanical insufflation-exsufflation (MIE), coupled with hypertonic saline (HS), may improve efficacy airway clearance and reduce risk of the maneuver. However, safety of MIE and HS in intubated patients have not been studied appropriately, which justifies a randomized evaluation compared to conventional secretion suctioning.

DETAILED DESCRIPTION:
Secretion suctioning (SS) in patients with artificial airway is a mandatory procedure, although occasionally painful, not tolerated and even causing traumatic injury to the respiratory mucosa.

Mechanical insufflation-exsufflation (MIE) and nebulized hypertonic saline with hyaluronic acid (HS-HA) have shown efficacy and safety in patients with chronic neuromuscular and pulmonary diseases, achieving aspiration and fluidification of respiratory secretions, respectively, as well as good tolerance.

Only anecdotal experience about the safety of MIE and HS-HA in critically ill patients with artificial airway and mechanical ventilation is available.

Background: Both MIE and HS-HA facilitate the drainage of secretions from the distal airway (compared to conventional catheter suctioning, the effect of which is supposed to be limited to the trachea) Both measures may prove to be efficacious in the prevention (through airway clearance of secretions) and concomitant treatment (reduction of inoculum or "draining the lung") of lower respiratory tract infections (tracheobronchitis and pneumonia).

ELIGIBILITY:
Inclusion Criteria:

* Artificial airway ( endotracheal tube or tracheostomy cannula) with pressure cuff.
* Need for aspiration of secretions
* Informed consent

Exclusion Criteria:

* Macroscopic hemoptysis.
* Acute bronchospasm
* Uncrontrolled muscular contractions, like tremor, myoclonus or other.
* Confirmed pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Aggregate cardiovascular and respiratory adverse events of mechanical insufflation-exsufflation and hypertonic saline. | 1 hour
  Comparative incidence of aggregate hemodynamic and respiratory adverse events.
  Adverse events criteria are predefined and will be expressed as:
  * Percentage of patients meeting aggregate predefined hemodynamic or respiratory adverse event criteria per study group.
  * Percentage of specific predefined adverse events (outcome variable "yes" or "no"): Desaturation (pulse-oximetry, >5%), hemoptisis (yes or no), bronchospasm (needing bronchodilator therapy), pneumothorax (as assessed by chest X-ray), hypotension (>30% or >10% increase in noradrenaline infusion from baseline), hypertension (>30% or >10% decrease in noradrenaline infusion from baseline), tachycardia (>90 bpm or >30% increase), bradycardia (<40 bpm), arrythmias (supra ventricular, requiring therapy), atelectasis (as assessed by chest X-ray), and other complications occuring during or within 1 hour after the procedure.
Pain score during mechanical insufflation-exsufflation and hypertonic saline as assessed by quantitative a pain scoring systems. | 1 hour
  Comparative pain scores of the study procedures in the 4 study groups will be assessed using the "ESCID" pain score (EScala de Conductas Indicadoras de Dolor, ranging from 0, no pain, to >6, intense pain, see citations) at baseline, during the procedure and at 5 and 60 minutes after the aspiration of respiratory secretions.
  Both comparison of the score at the 4 study time-points and their variations between time-points will be analysed.
Sedation/agitation score during mechanical insufflation-exsufflation and hypertonic saline as assessed by a quantitative sedation/agitation system. | 1 hour
  Comparative sedation/agitation score of the study procedures in the 4 study groups will be assessed using the RASS (Richmond Agitation-Sedation Scale, see citations), range -5, un-arousable, to +5, combative) at baseline, during the procedure and at 5 and 60 minutes after the aspiration of respiratory secretions.
Sedation/responsiveness score during mechanical insufflation-exsufflation and hypertonic saline as assessed by quantitative a sedation scoring system. | 1 hour
  Comparative sedation/responsiveness score of the study procedures in the 4 study groups will be assessed using the responsiveness "Ramsay" Sedation Scale, range from 1, anxious and agitated, to 6, no response to stimulus, see citations) at baseline, during the procedure and at 5 and 60 minutes after the aspiration of respiratory secretions.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Sanchez Garcia, MD, PhD, Principal Investigator — Hospital Clinico San Carlos
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain

REFERENCES:
- [Background] Latorre-Marco I, Acevedo-Nuevo M, Solis-Munoz M, Hernandez-Sanchez L, Lopez-Lopez C, Sanchez-Sanchez MM, Wojtysiak-Wojcicka M, de Las Pozas-Abril J, Robleda-Font G, Frade-Mera MJ, De Blas-Garcia R, Gorgolas-Ortiz C, De la Figuera-Bayon J, Cavia-Garcia C. Psychometric validation of the behavioral indicators of pain scale for the assessment of pain in mechanically ventilated and unable to self-report critical care patients. Med Intensiva. 2016 Nov;40(8):463-473. doi: 10.1016/j.medin.2016.06.004. Epub 2016 Aug 31. English, Spanish. PMID 27590592
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxalone-alphadolone. Br Med J. 1974 Jun 22;2(5920):656-9. doi: 10.1136/bmj.2.5920.656. PMID 4835444